CLINICAL TRIAL: NCT04272944
Title: Phase I Clinical Trial on the Tolerability and Pharmacokinetics of Recombinant Humanized Anti-PD-L1 Monoclonal Antibody MSB2311 Injection in the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Study of MSB2311 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Transcenta Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MSB2311-CSP-002
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: MSB2311 IV at 10 mg/kg Q2W, 20 mg/kg 3QW
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10 mg/kg Q2W (Experimental): 10 mg/kg IV every 2 weeks
  Interventions: Drug: 10 mg/kg Q2W
- 20 mg/kg Q3W (Experimental): 20 mg/kg IV every 3weeks
  Interventions: Drug: 20 mg/kg Q3W

INTERVENTIONS:
Drug: 10 mg/kg Q2W — 10 mg/kg MSB2311 every two weeks
  Other Names: MSB2311 10 Q2W
  Arms: 10 mg/kg Q2W
Drug: 20 mg/kg Q3W — 20 mg/kg MSB2311 every three weeks.
  Other Names: MSB2311 20 Q3W
  Arms: 20 mg/kg Q3W

SUMMARY:
This is a first-in-human (FIH), open-label, Phase 1 dose-Escalation Study of MSB2311, a humanized anti-PD-L1 monoclonal antibody, in subjects with advanced solid tumors. Qualified subjects will be enrolled to receive their assigned dose regimen of MSB2311 until disease progression or intolerable toxicity, withdrawal of consent, or end of study, whichever occurs first. The maximum treatment duration is 2 years. During the study, subjects will be evaluated for safety and toxicity, PK/PD, immunogenicity and anti-tumor activity of MSB2311.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary informed consent, knowledge of the study and willingness to follow and has ability to complete all trial procedures
* There is a histologically or cytologically confirmed, locally advanced or metastatic tumor that is not resectable

  * b period participants shall provide the archive paraffin embedding tumor tissue samples
* The eastern United States cooperative tumor group (ECOG) score was 0 or 1
* Expect to survive at least 3 months
* Subjects must have measurable lesions (at least 1 lesion) and minimum tumor-specific antigen levels where applicable
* If you have received antitumor therapy, you need to meet certain conditions
* There are suitable organs and hematopoietic functions
* Male subjects and female subjects of child-bearing age shall agree to take effective, investigator-approved contraceptive measures from the date of signing the informed consent until 3 months after the last administration

Exclusion Criteria:

* The patient has had a malignant tumor other than the tumor treated in this study within 5 years prior to the first administration, unless the medical examiner of the study group and sponsor agrees that the old tumor has been cured or will not metastasise or cause death in this study
* Adverse reactions to previous treatments did not return to CTCAE v4.03 rating ≤ 1, except for residual alopecia effect
* Patients who had been treated with anti-pd-1 or pd-l1 antibodies, or who had been treated with antibodies/drugs that target any other t-cell co-regulatory proteins within 12 weeks of the first administration of the drug in this study
* Patients with primary CNS tumors or CNS metastases known or identified during screening
* Subjects with active or pre-existing autoimmune disease that may recur or patients at high risk
* Patients who had major surgery in the first 4 weeks of screening and who were expected to have major surgery during the study period including a 28-day screening period
* Subjects who require systemic treatment with corticosteroids or other immunosuppressive drugs within 14 days prior to enrollment or during the study period
* Sudden pulmonary disease, interstitial pulmonary disease or pneumonia, or other uncontrolled systemic disease, including diabetes, pulmonary fibrosis, acute pulmonary disease, cardiovascular disease, including hypertension, except local interstitial pneumonia induced by radiotherapy
* A history of human immunodeficiency virus infection, or other acquired or congenital immunodeficiency, or a history of organ transplantation, or stem cell transplantation
* Had a history of tuberculosis, or had tuberculosis disease at the time of screening
* Patients with chronic hepatitis b or active hepatitis c.Hepatitis b carriers, stable hepatitis b after drug treatment and cured hepatitis c patients can be included in the group
* Patients who have been seriously infected within 4 weeks prior to first administration, or who have developed signs or symptoms of any active infection within the previous 2 weeks, or who require antibiotic treatment within the previous 2 weeks;Unexplained fever occurred before the first administration and the body temperature exceeded 38.5℃
* Subjects who have previously been known to have a severe allergic reaction to a macromolecular protein preparation/monoclonal antibody or to any component of the test drug
* Immune-related adverse events (irAE) grade ≥3 occurred after receiving immunotherapy
* Participated in clinical trials of other drugs within 4 weeks before enrollment
* A history of alcohol, drug or substance abuse within the last 1 year
* Has a clear history of neurological or psychiatric disorders, such as epilepsy, dementia, poor compliance
* A woman who is pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MSB2311 | Up to 90 days following the last dose
  Measured by number adverse events that are related to treatment
Maximum tolerated dose(MTD) or recommended phase2 dose（RP2D） | Up to 90 days following the last dose
  Measured by number of subjects experiencing DLT in each escalation cohort

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) for MSB2311 | Up to 30 days following the last dose
  Changes in AUC over time in subjects with MSB2311
Peak Plasma concentration (Cmax)for MSB2311 | Up to 30 days following the last dose
  Cmax is the maximum observed plasma concentration
Time to the Maximum Observed Plasma Concentration (Tmax) | Up to 30 days following the last dose
  Tmax is the time in hours/days to reach Cmax following dosing
Terminal elimination half-life (t1/2) | Up to 30 days following the last dose
  The time required for the plasma level of the study drug to decrease by one-half during the terminal elimination phase
Objective response rate (ORR) as measured by RESISTv1.1 | Up to 90 days following the last dose
Duration of response (DOR) as measured by RESISTv1.1 | Up to 90 days following the last dose
Progression-free survival (PFS) as measured by RESISTv1.1 | Up to 90 days following the last dose
Best overall response as measured by RESISTv1.1 | Up to 90 days following the last dose
Overall survival (OS) as measured by RESISTv1.1 | Up to 90 days following the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Mengde Wang, Study Director — Suzhou Transcenta Therapeutics Co., Ltd.
Locations (1):
- Mabspace Biosciences (Suzhou) Co., Ltd., Suzhou, Jiangsu, China